CLINICAL TRIAL: NCT01429077
Title: Augmenting Language Therapy for Aphasia: A Randomized Double-Blind Placebo-Controlled Trial of Levodopa in Combination With Speech-Language Therapy
Brief Title: Augmenting Language Therapy for Aphasia: Levodopa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leora Cherney, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H133G070074
Record Dates: First submitted 2011-08-02; First posted 2011-09-05 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Nonfluent Aphasia; Stroke
Keywords: Levodopa; Ischemic Stroke; Aphasia; Speech Rehabilitation
MeSH Terms: conditions — Aphasia, Broca; Stroke; Ischemic Stroke; Aphasia | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levodopa/carbidopa (Active Comparator): The study drug (100 mg levodopa / 25 mg carbidopa), is received orally 30-45 minutes before 1 hour of speech-language treatment, five days a week, for six weeks.
  Interventions: Drug: levodopa/carbidopa
- Inactive pill (Placebo Comparator): The placebo comparator (inactive pill) is received orally 30-45 minutes before 1 hour of speech-language treatment, five days a week, for six weeks.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: levodopa/carbidopa — The study drug (100 mg levodopa / 25 mg carbidopa), is received orally 30-45 minutes before 1 hour of speech-language treatment, five days a week, for six weeks.
  Other Names: Sinemet
  Arms: Levodopa/carbidopa
Drug: Placebo comparator — The placebo comparator (inactive pill) is received orally 30-45 minutes before 1 hour of speech-language treatment, five days a week, for six weeks.
  Arms: Inactive pill

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the medication levodopa, in combination with speech-language treatment, on the language outcome of study subjects with nonfluent aphasia (i.e. difficulty with the comprehension and expression of spoken and written language) following a stroke.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the most common cause of disability in the United States. According to the American Stroke Association, the prevalence of stroke in the U.S. is approximately 4.8 million with approximately 700,000 additional strokes occurring annually. Approximately 150,000 to 250,000 stroke survivors becoming severely and permanently disabled each year.

A common neurological deficit among stroke survivors, and thus a substantial contributor to post-stroke disability, is aphasia. The loss of, or difficulty with language is extremely debilitating and has enormous social and economic impact on quality of life. Presently, the only treatment available for persons with aphasia is speech-language rehabilitation.

With rehabilitation only, however, many patients achieve a less than satisfactory improvement in speech-language function, and thus are left with significant disability.

To enhance motor and language recovery in patients with neurological impairments, interest in the use of novel biological therapies, including pharmacological agents, has recently emerged. There is preliminary evidence that increased levels of dopamine, in combination with language treatment, may improve the deficits of aphasia following stroke. Most studies have investigated the adjunctive effects of the dopamine agonist bromocriptine, with mixed results. However, new evidence is suggesting that levodopa, a precursor to dopamine, may be more effective in promoting language learning.

This study proposes to evaluate the effectiveness of levodopa in study subjects with Broca's aphasia after stroke, delivered concurrent with speech-language rehabilitation.

The language changes in subjects who receive speech and language therapy combined with levodopa will be compared to that of subjects who receive the same speech-language rehabilitation but with a placebo (i.e. a pill that does not contain the study drug, levodopa). The two study groups will be compared to determine the degree to which improvements in language performance occur and the degree to which they are maintained over time.

The protocol is double-blind: neither subjects nor researchers will know whether a subject took levodopa or placebo until the study's conclusion.

ELIGIBILITY:
Inclusion Criteria:

* A single unilateral left-hemisphere stroke
* Nonfluent aphasia, with a mean length of utterance of 0-4 words and an Aphasia Quotient between 20 and 75 on the Western Aphasia Battery
* Age 21 or older.
* At least 6 months post-stroke
* Able to comply with the study protocol
* Premorbidly right-handed, as determined by the Edinburgh Handedness Inventory
* Fluent in English premorbidly
* Completed at least 8th grade education

Exclusion Criteria:

* More than one stroke
* Any other neurological condition that could potentially affect cognition or speech.
* Global aphasia or inability to participate in routine speech therapy.
* Major active psychiatric illness that may interfere with required study procedures.
* Untreated or inadequately treated depression.
* Has started taking a potentially confounding central nervous system (CNS) drug within the previous 2 months.
* Current abuse of alcohol or drugs
* Nursing a child or pregnant
* Participation in another drug, device or biologics trial within the preceding 90 days
* Unable to understand, cooperate or comply with study procedures
* Significant visual or auditory impairment
* History of sensitivity to ergot derivatives.
* Active medical illness or current medication that precludes safe participation in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Aphasia Research & Treatment, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Levodopa: The study drug (100 mg levodopa / 25 mg carbidopa), was received orally 30-45 minutes before 1 hour of speech-language treatment, five days a week, for six weeks.
- Inactive Pill: The inactive pill was received orally 30-45 minutes before 1 hour of speech-language treatment, five days a week, for six weeks.
Period: Overall Study
Arm/Group | Levodopa | Inactive Pill
Started | 19 | 17
Completed 6-week Intervention | 19 | 17
Completed | 19 | 14
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levodopa | Inactive Pill | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.8) | 52.6 (11.9) | 54.02 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Language Quotient (LQ) on the Western Aphasia Battery
Description: Includes a measure of auditory comprehension, oral expression, reading and written expression skills.
  The scale ranges from 1 - 100 with 100 being better. The change or gain score from baseline to immediately post-treatment (at 6 weeks) is reported. The larger the change score, the greater the improvement.
Time Frame: Change from Baseline in Western Aphasia Battery LQ at 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa/Carbidopa | Inactive Pill
Number analyzed (Participants) | 19 | 14
units on a scale | 3.16 (3.63) | 2.59 (3.41)

2. Secondary Outcome: Functional Communication Skills
Description: Scores derived from language sample analyses
Time Frame: Change from Baseline in functional communication skills at 6 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Participation in Everyday Activities
Description: Measures on CETI, QCL,BOSS, CCRSA.
Time Frame: Change from Baseline in participation in everyday activities at 6 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Western Aphasia Battery - Reading and Writing Scores
Time Frame: Change from Baseline in Western Aphasia Battery Reading and Writing scores at 6 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Western Aphasia Battery Aphasia Quotient (Maintenance)
Time Frame: Change in Western Aphasia Battery AQ from 6 weeks to 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Western Aphasia Battery Reading and Writing Scores (Maintenance)
Time Frame: Change in WAB Reading and Writing Skills from 6 weeks to 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Functional Communication Skills (Maintenance)
Time Frame: Change in functional communication skills from 6 weeks to 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Participation in Everyday Activities (Maintenance)
Time Frame: Change in participation in everyday activities from 6 weeks to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Levodopa | Inactive Pill
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 0/19 | 0/14

LIMITATIONS AND CAVEATS:
* Dosage and timing of the L-dopa in relation to the behavioral treatment may not have been optimum.
* Efficacy of the behavioral treatment in both arms may have overridden the enhancing effect of the l-dopa in one arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No